CLINICAL TRIAL: NCT00866411
Title: Outcomes of Cranial Electrotherapy Stimulation (CES) With Soldiers for Combat-Related Symptoms
Brief Title: Cranial Electrotherapy Stimulation (CES) for Soldiers With Combat-Related Symptoms
Acronym: CES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: LTC Mona O. Bingham, PhD, RN; Chief Nursing Reseach, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C.2007.147
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Last update posted 2009-03-20 (Estimated); Status verified 2009-03

CONDITIONS: Combat Related Symptoms; Irritability; Anger
Keywords: cranial electrotherapy stimulation; anxiety; depression; pain; sleep disturbance; combat exposure; post traumatic stress; health status; medication use; soldiers
MeSH Terms: conditions — Anxiety Disorders; Depression; Pain; Parasomnias

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: cranial electrotherapy stimulation (CES) with Alpha-Stim — three weeks of the cranial electrotherapy stimulation (CES) treatment (15 sessions of 60 minute treatments)
  Other Names: cranial electrotherapy stimulation; CES; Alpha-Stim; bioelectric medicine
Procedure: placebo — three weeks of placebo treatment via a double-blinded procedure so that neither the Soldier nor the study investigators will know whether the Soldier is receiving the actual treatment or placebo

SUMMARY:
The purpose of this double-blind randomized control research study is to determine if CES given in a group setting for soldiers experiencing irritability is effective to reduce the symptom of irritability.

ELIGIBILITY:
Inclusion Criteria:

* Soldiers over 18 years old or emancipated minors willing to sign an informed consent and complete all protocol requirements.
* Soldiers who score 4 or greater on the visual analog scale for irritability

Exclusion Criteria:

* Seizure disorders.
* Pregnancy. All female Soldiers will verify in the informed consent that they are not currently pregnant. Safety of stimulation has not been established during pregnancy and therefore we will exclude women who are or want to become pregnant during the course of the study.
* Concomitant therapy with an investigational drug or device, or participation in an investigational drug or device study within one month prior to entering this study
* Patients with a pacemaker or implanted defibrillator. The Alpha-Stim 100 may effect the operation of cardiac pacemakers (particularly demand type pacemakers) and therefore this population will be excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-05; Primary Completion 2009-05 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Irritability Visual Analog Scale | Baseline, daily x 3 weeks, 4 weeks

SECONDARY OUTCOMES:
State Anxiety Scale | Baseline, 3 weeks, 4 weeks
Pittsburgh Sleep Quality Index | Baseline, 3 weeks, 4 weeks
Epworth Sleepiness Scale | Baseline, 3 weeks, 4 weeks
General Sleep Disturbance Scale | Baseline, 3 weeks, 4 weeks
Sleep Self Care Questionnaire | Baseline, 3 weeks, 4 weeks
Combat Exposure Scale | Baseline
Trauma Imagery Scale | Baseline, 3 weeks, 4 weeks
State - Anxiety Scale | Baseline, 3 weeks, 4 weeks
Profile of Mood States | Baseline, 3 weeks, 4 weeks
Visual Analog | Daily x 3 weeks, 4 weeks
Center for Epidemiological Center for Epidemiological Studies - Depression Scale | Baseline, 3 weeks, 4 weeks
Depression Visual Analog | Daily x 3 weeks, 4 weeks
PTSD CheckList - Military Version | Baseline, 3 weeks, 4 weeks
Veteran's Outcomes Survey Short Form - 36 | Baseline, 3 weeks, 4 weeks
Medication Use Questionnaire | Baseline, 3 weeks, 4 weeks
Spielberger State-Trait Anger Expression Inventory-2(STAXI-2) | baseline, 3 weeks, 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mona O Bingham, PhD, Principal Investigator — Brooke Army Medical Center
Locations (2):
- United States (2):
  - Carl R. Darnall Army Medical Center, Fort Hood, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas